CLINICAL TRIAL: NCT06943898
Title: Investigation of the Acute Effects of Core Stabilization and 360-Degree Breathing Exercises on Balance and Proprioception in Individuals With Non-Specific Low Back Pain
Acronym: 360° Breath
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Selvin BALKİ, associate professor, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCU-FTR-SB-01
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Low Back Pain (LBP); Exercise; Core Stability
Keywords: core stability exercise; low back pain; exercise
MeSH Terms: conditions — Low Back Pain; Motor Activity | interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: two groups with a conventional therapy control group.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Core Exercises) (Other): Core Exercises Group
  Interventions: Other: Core Egzercise
- Intervention Group (Core Exercises + Breathing Exercises): (Other): Core Exercises + Breathing Exercises
  Interventions: Other: Core Exercises + Breathing Exercises

INTERVENTIONS:
Other: Core Egzercise — The core exercise group will perform core stabilization exercises for a total of 15 sessions, five days a week for three weeks. Exercises will include pelvic tilt, bridge, dead bug, bird dog, mini squats on a balance board, and wall planks. The number of repetitions will be increased from 10 to 20, and plank duration will be increased from 30 seconds to 45 seconds. A 5-minute warm-up and cool-down session will be included.
  Arms: Control Group (Core Exercises)
Other: Core Exercises + Breathing Exercises — This group will perform core stabilization exercises combined with the 360-degree breathing technique, for a total of 15 sessions over three weeks (five days a week).
  "360-degree breathing" is a novel breathing method targeting deep and controlled inhalations into various regions of the body. Unlike traditional breathing exercises, 360-degree breathing ensures that all directions of the lungs are equally ventilated.
  Arms: Intervention Group (Core Exercises + Breathing Exercises):

SUMMARY:
This study is designed as a single-blind randomized controlled trial. Male and female patients aged 18-65 years with complaints of non-specific low back pain (NSLBP) lasting longer than 12 weeks will be included in the study. Participants will be randomly assigned into two parallel groups: control and intervention. The control group will perform core stabilization exercises five days a week for three weeks. In the intervention group, core stabilization exercises will be combined with 360-degree breathing exercises. To our knowledge, there is no randomized controlled trial investigating the effect of combining core stabilization with 360-degree breathing in individuals with NSLBP. The aim of this study is to examine the acute effects of combining 360-degree breathing techniques with core stabilization exercises on balance and proprioception in individuals with NSLBP.

DETAILED DESCRIPTION:
Low back pain is a major health problem worldwide. Non-specific low back pain (NSLBP) is the most common form of back pain. The lifetime prevalence of back pain can reach up to 84%. Various non-pharmacological and non-invasive methods are used for back pain management. One such method is core stabilization exercises. Core stabilization exercises enhance trunk stability by activating the muscles around the spine and have the potential to improve balance in individuals with NSLBP. This may help overcome balance disorders associated with pain and contribute to safer movements in daily life activities. Breathing exercises, by activating the diaphragm muscle, support spinal stability and provide benefits in pain management. It is known that breathing supports trunk stability through its relationship with core muscles and strengthens balance mechanisms. Studies in this field show that stabilization exercises can provide short-term improvements, especially in balance. However, the combined effects of core stabilization and breathing exercises in individuals with NSLBP have not been fully investigated. Therefore, this study aims to investigate the acute effects of combining 360-degree breathing exercises with core stabilization exercises on balance and proprioception in individuals with NSLBP.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain persisting for at least 3 months
* No neurological, rheumatological, or musculoskeletal system problems

Exclusion Criteria:

* Individuals with neurological, vestibular, or serious orthopedic conditions that may cause physical disability
* Patients with back-leg or dorsolumbar pain due to lumbar disc protrusion or fracture
* Cancer patients
* Individuals with acute infections
* Individuals with respiratory system diseases
* Individuals with any mental disorder that would prevent participation in the study assessment
* Pregnant individuals

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
• Proprioception Assessment | 3 week
  Proprioception will be evaluated using an inclinometric method. An inclinometer is usually placed and fixed at the L3-L4 segment of the lumbar spine. The patient will be asked to achieve and then reproduce a target position. The difference between the reference angle and the reproduced angle (position error) will be recorded as a measure of proprioceptive perception.
Y Balance Test (YBT) | 3 week
  The Y Balance Test (YBT) will be used to assess balance. Patients will remove their shoes and place the stance foot on the center footplate of the YBT platform. They will attempt to reach maximally with the opposite leg in three directions (anterior, posteromedial, and posterolateral), maintaining balance on the stance leg. Maximum reach distances will be recorded.

SECONDARY OUTCOMES:
Core Muscle Endurance Assessment: | 3 week
  Core endurance will be assessed using McGill's protocol, including trunk extension, trunk flexion, lateral bridge, and prone bridge tests.
  1. Trunk Extension Test:
     In the prone position, the trunk is extended off the edge of the table to the level of the anterior superior iliac spine. Upper body is supported by arms on a chair, hips and legs are fixed. After removing the support, the individual crosses their arms over the chest. The time the individual can hold this position is recorded in seconds.
  2. Trunk Flexion Test:
     The patient sits on the table with hips and knees at 90° flexion and the trunk at 60° flexion. Feet are secured to the table, arms crossed over the chest. After removing the back support, the individual maintains the position as long as possible. Time is recorded in seconds.
  3. Lateral Bridge Test:
  The patient lies in a side-lying position with the lower arm flexed at 90° and forearm on the table. The upper arm is crossed over the chest. Lower extremities are extended
Visual Analog Scale (VAS) | 3 week
  Pain levels will be evaluated using the Visual Analog Scale (VAS), ranging from 0 to 10. A score of 0 indicates no pain; 1-4 indicates mild pain; 5-6 indicates moderate pain; 7-10 indicates severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Balki, PhD, Study Director — Sivas Cumhuriyet University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation
Locations (1):
- Sivas Cumhuriyet University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation, Sivas, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No